CLINICAL TRIAL: NCT05141396
Title: Implementation of Coordinated Spontaneous Awakening and Breathing Trials Using Telehealth-Enabled, Real-Time Audit and Feedback for Clinician Adherence: A Type II Hybrid Effectiveness-Implementation
Brief Title: Telehealth-Enabled, Real-time Audit and Feedback for Clinician AdHerence (TEACH)
Acronym: TEACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1051681; U01HL159878 (NIH)
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Respiration, Artificial
Keywords: Invasive Mechanical Ventilation; Coordinated Spontaneous Awakening and Breathing Trials
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Telehealth- enabled support plus usual audit and feedback for SAT/SBT adherence (Experimental): Usual audit and feedback + telehealth-enabled support
  Interventions: Other: Telehealth- enabled support for SAT/SBT adherence; Other: Usual audit and feedback for SAT/SBT adherence
- Control - Usual audit/feedback for SAT/SBT adherence only (Active Comparator): Usual audit and feedback
  Interventions: Other: Usual audit and feedback for SAT/SBT adherence

INTERVENTIONS:
Other: Telehealth- enabled support for SAT/SBT adherence — Telehealth-enabled support over and above usual audit and feedback includes identifying candidates for spontaneous awakening and breathing trials, prompting bedside providers and guiding execution of the coordinated spontaneous awakening and breathing trials as needed.
  Arms: Intervention - Telehealth- enabled support plus usual audit and feedback for SAT/SBT adherence
Other: Usual audit and feedback for SAT/SBT adherence — Usual audit and feedback

SUMMARY:
The purpose of this trial is to evaluate if augmenting a usual audit and feedback implementation approach with telehealth-enabled support improves coordinated spontaneous awakening/breathing trials and patient outcomes for mechanically ventilated patients.

DETAILED DESCRIPTION:
Sedation and analgesia are utilized with invasive mechanical ventilation (IMV) to improve patient comfort and synchrony with the mechanical ventilator. Prolonged sedation, however, may result in increased time on IMV and increased risk for ventilator associated pneumonia, delirium, and poor long-term cognitive outcomes. Daily interruptions in sedation [spontaneous awakening trials (SAT)] coordinated with daily spontaneous breathing trials (SBT) reduce mortality, increase ventilator free days, decrease intensive care unit (ICU) length of stay, and reduces ventilator-associated events. Coordination of spontaneous awakening and breathing trials (C-SAT/SBT), however, are underutilized due to significant barriers to implementation and adherence. This cluster-randomized hybrid implementation/effectiveness trial will compare C-SAT/SBT adherence and clinical outcomes in the presence of traditional audit and feedback implementation strategies alone or augmented with a novel Telehealth-Enabled, real-time Audit and feedback for Clinician adHerence ("TEACH") implementation strategy.

ELIGIBILITY:
Inclusion criteria:

* Patient age >=16 years admitted to study hospital ICU
* Intubated and mechanically ventilated

Exclusion criteria:

* Patient with pre-existing brain death admitted to study hospital for organ donation
* Died within 24 hours of intubation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13400 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Adherence to C-SAT/SBT | intubation to extubation - an average of 5 days
  Fraction of eligible days on which coordinated spontaneous awakening trial and spontaneous breathing trial completed.
Ventilator-free days to day 28 | 28 days
  ventilator-free days to day 28

SECONDARY OUTCOMES:
30-day Mortality | 30 days
Hospital Length of Stay | Through hospital discharge, an average of 10 days
90-day Mortality | 90 Days
New ventilator-associated pneumonia | Through hospital discharge, an average of 10 days
ICU Length of Stay | Through hospital discharge, an average of 10 days
Reintubation | intubation to extubation - an average of 5 days
Unintentional Extubation | intubation to extubation - an average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Colin Grissom, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (11):
- United States (11):
  - American Fork Hospital, American Fork, Utah
  - Cedar City Hospital, Cedar City, Utah
  - Layton Hospital, Layton, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - Mckay Dee Hospital, Ogden, Utah
  - Utah Valley Hospital, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Alta View Hospital, Sandy City, Utah
  - St. George Regional Hospital, St. George, Utah

IPD SHARING:
Plan to Share IPD: Yes
In order to protect patient privacy and comply with relevant regulations, identified data will be unavailable. Requests for deidentified data from qualified researchers with appropriate ethics board approvals and relevant data use agreements will be processed by the Intermountain Office of Research, officeofresearch@imail.org.

REFERENCES:
- [Derived] Grissom CK, Holubkov R, Carpenter L, Hanna B, Jacobs JR, Jones C, Knighton AJ, Leither L, Lisonbee D, Peltan ID, Winberg C, Wolfe D, Srivastava R. Implementation of coordinated spontaneous awakening and breathing trials using telehealth-enabled, real-time audit and feedback for clinician adherence (TEACH): a type II hybrid effectiveness-implementation cluster-randomized trial. Implement Sci. 2023 Sep 21;18(1):45. doi: 10.1186/s13012-023-01303-1. PMID 37735443